CLINICAL TRIAL: NCT02733614
Title: A Proof of Concept (POC) Clinical Trial for Post-Traumatic Stress Disorder (PTSD) With a First-In-Class Vasopressin 1a Receptor Antagonist (SRX246)
Brief Title: Proof-of-concept Study to Assess the Efficacy and Safety of SRX246 in Adults With PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: Azevan Pharmaceuticals (Industry)
Collaborators: Weill Medical College of Cornell University (Other); United States Department of Defense (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN010
Record Dates: First submitted 2016-03-29; First posted 2016-04-11 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — SRX246

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SRX246 (Experimental): SRX246 160 mg BID, oral administration, capsules, daily for 8 weeks
  Interventions: Drug: SRX246
- Placebo (Placebo Comparator): oral administration, capsules, daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SRX246 — novel V1a receptor antagonist
  Arms: SRX246
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
18-week, crossover, double-blind, randomized, placebo controlled proof-of-concept study to assess the efficacy and safety of SRX246 (160 mg bid) vs placebo in 52 adult veterans and civilians with a primary diagnosis of PTSD. Subjects will be randomly assigned in a double-blind fashion to 2 groups in a crossover design. The first group will receive SRX246 for 8 weeks followed by 8 weeks of placebo, while the second group will receive placebo for 8 weeks followed by 8 weeks of SRX246. Both groups will engage in a 7-day washout period between treatments. Subjects will be assessed at baseline and then every 2 weeks during the trial using the CAPS.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable, current diagnosis of PTSD

Exclusion Criteria:

* Medically unstable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Assessment of overall clinical improvement | 18 weeks
  Measured using the Clinician Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 18 weeks
  Assessments of adverse events (AEs), dose reductions and dropouts due to AEs
Reduction in depressive symptoms | 18 weeks
  Measured using the Beck Depression Inventory (BDI)
Reduction in anger and aggression | 18 weeks
  Measured using the Overt Aggression Scale-Modified (OAS-M)
Reduction in irritability | 18 weeks
  Measured using the Sheehan Irritability Scale (SIS)
Improvement in overall functioning | 18 weeks
  Measured using the Medical Outcomes Study Short-Form 12-Item Health Survey (SF-12)
Improvement in quality of life | 18 weeks
  Measured using the Sheehan Disability Scale (SDS)
Improvement in sleep quality | 18 weeks
  Measured using the Pittsburgh Sleep Quality Index (PSQI)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No